CLINICAL TRIAL: NCT05516602
Title: Improving HIV Prevention Among Adolescent Girls and Young Women (AGYW) in Uganda
Acronym: Peers for PREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Collaborators: Uganda Virus Research Institute (UVRI) (Unknown); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RGYM220701
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: HIV-1-infection
Keywords: Adolescent Girls and Young Women; Oral PrEP; Peer Support; Uganda

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer Support (Experimental): Standard health worker counselling during clinic visits plus peer support over the weekends.
  Interventions: Other: Peer Support
- Standard (No Intervention): Standard health worker counselling during clinic visits.

INTERVENTIONS:
Other: Peer Support — Peer-led support groups over the weekend will include the following activities:
  * Peer leader counselling on oral PrEP and HIV risk reduction
  * Peer leader discussion to dispel myths and misconceptions around oral PrEP
  * Peer leader sharing of experiences of daily pill taking
  * Participants sharing experiences of influencers and barriers to oral PrEP uptake and adherence followed by a discussion by group members.
  * 1-2 role plays per support group session.
  Arms: Peer Support

SUMMARY:
Purpose: The purpose of the project is to evaluate a peer support intervention aimed at improving uptake of and adherence to oral PrEP.

Main Study Aim:

To evaluate a peer support intervention aimed at improving uptake of and adherence to oral pre-exposure prophylaxis (PrEP), and its effect on sexual behavioral and reproductive health outcomes

Study Objectives:

i. To evaluate the effect of a peer support intervention on uptake of and adherence to oral PrEP among 14-24-year-old AGYW at risk of HIV infection in Kampala, Uganda.

ii. To evaluate the effect of the peer support intervention aimed at improving oral PrEP uptake and adherence, on sexual behavior and reproductive health outcomes among AGYW in Kampala, Uganda.

Design An individually randomized controlled trial with parallel group design and 1:1 randomization in the intervention and control arms.

Population: 14-24-year old AGYW at risk of HIV infection in Kampala.

Control arm: Standard health worker counselling during clinic visits.

Intervention arm: Standard health worker counselling during clinic visits + peer support groups over the weekend.

DETAILED DESCRIPTION:
1 INTRODUCTION 1.1 Background Adolescent girls and young women (AGYW) aged 15-24 years in Sub-Saharan Africa (SSA) are at substantial risk for HIV infection and in 2020, AGYW accounted for 32% of new HIV infections in East and Southern Africa [1]. In the general population in Uganda, the HIV prevalence among AGYW is estimated at 1.8% among 15-19 year-olds and 5.1% among 20-24 year-olds [2]. The prevalence among AGYW living in fishing communities in Uganda, and young female sex workers (FSWs) is even higher estimated at 15.4% and 22.5% respectively [3, 4]. During recent years, biomedical interventions for HIV prevention have been developed and are currently at different stages of the pipeline with some already approved for use. For example, anti-retroviral (ARV) implants for pre-exposure prophylaxis (PrEP) to protect HIV negative girls from becoming HIV infected, have recently been assessed in pre-clinical studies [5, 6]. Other biomedical interventions for HIV prevention among vulnerable HIV negative sub-groups, including AGYW in SSA, have further been assessed in clinical trials for example: the Dapivirine vaginal ring (DVR) [7, 8], long acting injectable PrEP [9, 10], HIV vaccines [11] and oral PrEP [12, 13]. Oral PrEP is a single pill taken once daily during periods of risk to HIV infection, and is highly efficacious when adherence is good (>90%) [12]. Tenofovir is one of the most common HIV drugs and tenofovir-based oral PrEP is also one of the World Health Organization (WHO) approved biomedical HIV prevention interventions [14, 15]. In 2016, the Uganda government approved use of oral PrEP for HIV prevention among individuals at substantial risk of HIV infection [16], and increased access to targeted key populations including AGYW. The HIV prevention landscape is promising as other novel biomedical HIV prevention interventions are in various stages of development, including long acting injectable PrEP, anti-retroviral (ARV) implants and HIV vaccines. The Dapivirine vaginal ring is approved by WHO as an additional HIV prevention choice for women [17], has been approved for use in South Africa [18] and, has been added to the drug register of the National Drug Authority in Uganda [19]. Injectable cabotegravir may also be available soon having shown efficacy in the HIV Prevention Trials Network (HPTN084) study [10]. End-user preferences for HIV prevention products may predict method uptake [20] and there is a need to increase researchers' knowledge about current preferences for HIV prophylaxis among AGYW in SSA who continue to be at substantial risk of HIV.

1.2 Oral PrEP Uptake and Adherence among Adolescent Girls and Young Women Oral PrEP is still currently the only available biomedical HIV prevention method in most parts of SSA. PrEP implementation projects have been facilitated through the U.S. President's Emergency Plan for AIDS Relief (PEPFAR) funding. Despite the potential benefits in HIV prevention, uptake and adherence to oral PrEP remain low among AGYW in Uganda and other parts of SSA [21, 22]. A recent study among AGYW in Kampala, Uganda, with high reported prevalence of being engaged in sex for compensation, also found a low oral PrEP uptake (31%) in this population [23]. The study also found that the uptake was higher in respondents with more sexual partners and among those who showed higher preference for oral PrEP over other biomedical HIV prevention methods when asked at enrolment. Importantly, tests for Tenofovir levels in blood showed very low adherence. Conversely, the Prevention Options for Women Evaluation Research (POWER) project which also enrolled 16-25-year-old AGYW in Kenya and South Africa reported high PrEP uptake (90%) associated with higher risk behavior, intimate partner violence (IPV), depression and chlamydia/ gonorrhea diagnosis [24]. Despite high PrEP uptake, the POWER project reported early discontinuation of PrEP use due to side effects, challenges with accessing services and product characteristics such as need for daily dosing [24, 25]. Other studies have identified pill burden, side effects [21, 22], low risk perception [26, 27] and limited awareness of oral PrEP [28] as barriers to PrEP uptake among AGYW in SSA. Interviews with potential PrEP users in multiple settings in central Uganda also showed that stigma, transport costs to get PrEP refills, accessibility, busy schedules, and forgetfulness were barriers to PrEP uptake while closeness of PrEP providers to one's home was a facilitator [29]. Thus, there is a need for interventions that may promote PrEP use among AGYW populations in SSA who are at increased risk of HIV infection.

1.3 Rationale Peer-to-peer support is one of the strategies proposed for improving HIV prevention and promotion of safer sexual behaviors in the Uganda National HIV research agenda [30], but there is limited evidence of its effectiveness in PrEP programs. Studies show that young people easily take on behaviors when in groups than as individuals, easily adopt behaviors and norms of their peers [31, 32], and are more easily affected by peer influence compared to children and older adults [33]. Among young people living with HIV in Zimbabwe, peer-led psycho-social support services among HIV positive individuals led to a 13% decrease in detectable viremia at 6 months compared with counselling delivered by health care workers (HCWs) [34]. A recent study among refugee adolescents in Northern Uganda showed same day acceptance of contraception was 9% higher among those who received peer counselling compared to counselling provided by HCWs [35]. In addition, trained peers have led to improvements in the HIV care and treatment cascade and contraceptive use through peer counselling, peer support for example delivery of interventions, peer referral etc. [36, 37]. Previous evidence suggests that peer counselling and support interventions have improved HIV testing, utilization of health care services, anti-retroviral therapy (ART) initiation, adherence to treatment, adherence to HIV viral load testing at 6 months and HIV viral suppression among young people living with HIV in Zimbabwe [37, 38]. Peer support interventions may therefore also improve oral PrEP uptake and adherence, and also reduce sexual behavior risk among AGYW, but this has not been widely studied.

2. STUDY AIMS AND RESEARCH QUESTIONS 2.1 The main aim of this project is to evaluate the effect of a peer support intervention on oral PrEP uptake and adherence, sexual behavioral and reproductive health outcomes of 14-24-year-old AGYW who are at high risk of HIV infection.

2.2 Research Questions i. What is the effect of a peer support intervention on uptake of and adherence to oral PrEP among AGYW aged 14-24 years at high risk of HIV infection in Uganda? ii. What are the effects of a peer support intervention for oral PrEP uptake and adherence on sexual behavior and reproductive health outcomes of AGYW aged 14-24 years at high risk of HIV infection in Uganda?

The investigators hypothesize that the peer support intervention will: (i) improve oral PrEP uptake and adherence among AGYW; (ii) reduce sexual behavioral risk, pregnancy and sexually transmitted infection (STI) rates

ELIGIBILITY:
Inclusion Criteria:

* HIV negative (assessed through rapid blood test)
* Sexually active in the past 3 months
* 14-24 years
* Hepatitis B negative for those who initiate oral PrEP
* Willing to undergo study procedures

Exclusion Criteria:

* HIV infection
* Currently taking oral PrEP
* Known allergy to common medications, components of oral PrEP or contraceptives
* Pregnant
* An acute or chronic illness that may affect volunteer participation or achieving study objectives
* A condition or situation that in the opinion of the PI/designee would preclude provision of informed consent, or otherwise interfere with achieving the study objectives

Ages: 14 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 394 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
The proportion of enrolled participants who take up oral PrEP after randomization to peer support or the standard | Measured from enrolment to the end of follow up at 12 months
  Number of participants who take up oral PrEP divided by the total number enrolled. PrEP uptake was measured as a participants accepting the offer of oral PrEP and picking their first month's supply from the clinic.
The proportion of volunteers who take up oral PrEP and adhere to oral PrEP after randomization to peer support or the standard | 3 monthly measurements from enrolment to the end of follow up at 12 months
  Number of participants who adhere to oral PrEP divided by the total number taking oral PrEP. Adherence was measured using self reports, pill counts and rapid urine tenofovir kits
Time in days to oral PrEP uptake from the date it is offered after randomization to peer support or the standard. | Measured from enrolment to the end of follow up at 12 months
  Number of days from the date a participant is offered oral PrEP to the date they pick the first month's supply from the clinic.

SECONDARY OUTCOMES:
Total number of sexual partners in the past 3 months in the peer support group compared to the standard | 3 monthly measurements from enrolment to the end of follow up at 12 months
  Proportion of participants having a specific risk score for total sexual partners in the past 3 months comparing the peer support group and the standard. Risk scores 1-4 assigned for number of sexual partners in the past 3 months as follows:
  * 0= no sexual partners
  * 1= 1 sexual partner
  * 2= 2-4 sexual partners
  * 3= 5-9 sexual partners
  * 4= ≥10 sexual partners
STI and pregnancy incidence at follow up in the peer support group compared to the standard | 3 monthly measurements from enrolment to the end of follow up at 12 months
  The number of new STI infections and pregnancies recorded every 3 months in the peer support group compared to the standard.
  Having an incident STI (Yes/ No) defined as the first new diagnosis of chlamydia and/ or gonorrhoea (positive urine GeneXpert) in a participant who tested negative for either STI (negative urine GeneXpert) at enrolment.
  Having an incident pregnancy (Yes/ No) defined as the first new pregnancy (positive urine βHCG) in a participant who was not pregnant (negative urine βHCG ) at enrolment.
Condom use with total sexual partners in the past 3 months in the peer support groups compared to the control | 3 monthly measurements from enrolment to study end at 12 months
  Proportion of participants with a specific risk score for reported condom use with total sexual partners in the past 3 months comparing the peer support groups and the control. Risk scores assigned for reported condom use with sexual partners in the past 3 months as follows:
  * 1= used condoms always
  * 2= used condoms most times
  * 3= used condoms sometimes
  * 4= did not use condoms at all
The proportion of participants who are not using a modern contraceptive at baseline and take up a modern contraceptive method at any time during the study | 3 monthly measurements from enrolment to the end of follow up at 12 months
  Number of participants who take up a modern contraceptive method during the study.
  Contraceptive uptake (Yes/ No) defined as a participant who reported not using contraception at enrolment taking up a contraceptive method at any time during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yunia Mayanja, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- MRC/UVRI and LSHTM, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: No
Data sharing will follow the MRC/UVRI and LSHTM Unit policies and the General Data Protection Regulation (GDPR). Before data is shared, data sharing agreements will be agreed and signed by the responsible parties ensuring participant confidentiality is kept. All personal data/ identifiers will be anonymized before sharing so that records cannot be linked back to an individual. Data will be shared through protected links and servers and not by emails.

REFERENCES:
- [Background] UNAIDS Fact Sheet, Global HIV Statistics. 2021.
- [Background] Ministry of Health, Uganda Population-based HIV Impact Assessment (UPHIA) 2016-2017: Final Report. Kampala: Ministry of Health; July, 2019. 2019.
- [Background] Nanyonjo G, Asiki G, Ssetaala A, Nakaweesa T, Wambuzi M, Nanvubya A, Mpendo J, Okech B, Kitandwe PK, Nielsen L, Nalutaaya A, Welsh S, Bagaya BS, Chinyenze K, Fast P, Price M, Kiwanuka N. Prevalence and correlates of HIV infection among adolescents and young people living in fishing populations along Lake Victoria Fishing Communities in Uganda. Pan Afr Med J. 2020 Nov 2;37:208. doi: 10.11604/pamj.2020.37.208.26124. eCollection 2020. PMID 33505576
- [Background] Swahn MH, Culbreth R, Salazar LF, Kasirye R, Seeley J. Prevalence of HIV and Associated Risks of Sex Work among Youth in the Slums of Kampala. AIDS Res Treat. 2016;2016:5360180. doi: 10.1155/2016/5360180. Epub 2016 Apr 28. PMID 27239340
- [Background] Nel A, van Niekerk N, Kapiga S, Bekker LG, Gama C, Gill K, Kamali A, Kotze P, Louw C, Mabude Z, Miti N, Kusemererwa S, Tempelman H, Carstens H, Devlin B, Isaacs M, Malherbe M, Mans W, Nuttall J, Russell M, Ntshele S, Smit M, Solai L, Spence P, Steytler J, Windle K, Borremans M, Resseler S, Van Roey J, Parys W, Vangeneugden T, Van Baelen B, Rosenberg Z; Ring Study Team. Safety and Efficacy of a Dapivirine Vaginal Ring for HIV Prevention in Women. N Engl J Med. 2016 Dec 1;375(22):2133-2143. doi: 10.1056/NEJMoa1602046. PMID 27959766
- [Background] Nel A, van Niekerk N, Van Baelen B, Malherbe M, Mans W, Carter A, Steytler J, van der Ryst E, Craig C, Louw C, Gwetu T, Mabude Z, Kotze P, Moraba R, Tempelman H, Gill K, Kusemererwa S, Bekker LG, Devlin B, Rosenberg Z; DREAM Study Team. Safety, adherence, and HIV-1 seroconversion among women using the dapivirine vaginal ring (DREAM): an open-label, extension study. Lancet HIV. 2021 Feb;8(2):e77-e86. doi: 10.1016/S2352-3018(20)30300-3. PMID 33539761
- [Background] Kirby T. Cabotegravir, a new option for PrEP. Lancet Infect Dis. 2020 Jul;20(7):781. doi: 10.1016/S1473-3099(20)30497-7. No abstract available. PMID 32592669
- [Background] Moretlwe, S.D., et al., Long acting injectable cabotegravir is safe and effective in preventing HIV infection in cisgender women: interim results from HPTN 084. Journal of the International AIDS Society
- [Background] Laher F, Bekker LG, Garrett N, Lazarus EM, Gray GE. Review of preventative HIV vaccine clinical trials in South Africa. Arch Virol. 2020 Nov;165(11):2439-2452. doi: 10.1007/s00705-020-04777-2. Epub 2020 Aug 14. PMID 32797338
- [Background] Baeten JM, Donnell D, Ndase P, Mugo NR, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kakia A, Odoyo J, Mucunguzi A, Nakku-Joloba E, Twesigye R, Ngure K, Apaka C, Tamooh H, Gabona F, Mujugira A, Panteleeff D, Thomas KK, Kidoguchi L, Krows M, Revall J, Morrison S, Haugen H, Emmanuel-Ogier M, Ondrejcek L, Coombs RW, Frenkel L, Hendrix C, Bumpus NN, Bangsberg D, Haberer JE, Stevens WS, Lingappa JR, Celum C; Partners PrEP Study Team. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. N Engl J Med. 2012 Aug 2;367(5):399-410. doi: 10.1056/NEJMoa1108524. Epub 2012 Jul 11. PMID 22784037
- [Background] Haberer JE, Baeten JM, Campbell J, Wangisi J, Katabira E, Ronald A, Tumwesigye E, Psaros C, Safren SA, Ware NC, Thomas KK, Donnell D, Krows M, Kidoguchi L, Celum C, Bangsberg DR. Adherence to antiretroviral prophylaxis for HIV prevention: a substudy cohort within a clinical trial of serodiscordant couples in East Africa. PLoS Med. 2013;10(9):e1001511. doi: 10.1371/journal.pmed.1001511. Epub 2013 Sep 10. PMID 24058300
- [Background] Guideline on When to Start Antiretroviral Therapy and on Pre-Exposure Prophylaxis for HIV. Geneva: World Health Organization; 2015 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK327115/ PMID 26598776
- [Background] World Health Organisation, WHO implementation tool for pre-exposure prophylaxis ( PrEP) of HIV infection: module 12: adolescents and young adults. 2018.
- [Background] Ministry of Health, Consolidated guidelines for the prevention and treatment of HIV and AIDS in Uganda. 2016.
- [Background] World Health Organisation, WHO recommends the dapivirine vaginal ring as a new choice for HIV prevention for women at substantial risk of HIV infection. 2021.
- [Background] Solai, L. and H. Seltzer, South Africa Approves Dapivirine Vaginal Ring for Use by Women. 2022.
- [Background] National Drug Authority, Drug Register. 2022.
- [Background] UNAIDS, Invest in HIV Prevention. 2015.
- [Background] Koss CA, Charlebois ED, Ayieko J, Kwarisiima D, Kabami J, Balzer LB, Atukunda M, Mwangwa F, Peng J, Mwinike Y, Owaraganise A, Chamie G, Jain V, Sang N, Olilo W, Brown LB, Marquez C, Zhang K, Ruel TD, Camlin CS, Rooney JF, Black D, Clark TD, Gandhi M, Cohen CR, Bukusi EA, Petersen ML, Kamya MR, Havlir DV; SEARCH Collaboration. Uptake, engagement, and adherence to pre-exposure prophylaxis offered after population HIV testing in rural Kenya and Uganda: 72-week interim analysis of observational data from the SEARCH study. Lancet HIV. 2020 Apr;7(4):e249-e261. doi: 10.1016/S2352-3018(19)30433-3. Epub 2020 Feb 19. PMID 32087152
- [Background] Mugwanya KK, Pintye J, Kinuthia J, Abuna F, Lagat H, Begnel ER, Dettinger JC, John-Stewart G, Baeten JM; PrEP Implementation for Young Women and Adolescents (PrIYA) Program. Integrating preexposure prophylaxis delivery in routine family planning clinics: A feasibility programmatic evaluation in Kenya. PLoS Med. 2019 Sep 3;16(9):e1002885. doi: 10.1371/journal.pmed.1002885. eCollection 2019 Sep. PMID 31479452
- [Background] Mayanja Y, Kamacooko O, Lunkuse JF, Muturi-Kioi V, Buzibye A, Omali D, Chinyenze K, Kuteesa M, Kaleebu P, Price MA. Oral pre-exposure prophylaxis preference, uptake, adherence and continuation among adolescent girls and young women in Kampala, Uganda: a prospective cohort study. J Int AIDS Soc. 2022 May;25(5):e25909. doi: 10.1002/jia2.25909. PMID 35543110
- [Background] Rousseau-Jemwa, E., et al. Early Persistence of HIV Pre-exposure Prophylaxis (PrEP) in African Adolescent Girls and Young Women (AGYW) from Kenya and South Africa. in HIV Research for Prevention. 2018.
- [Background] Celum CL, Delany-Moretlwe S, Baeten JM, van der Straten A, Hosek S, Bukusi EA, McConnell M, Barnabas RV, Bekker LG. HIV pre-exposure prophylaxis for adolescent girls and young women in Africa: from efficacy trials to delivery. J Int AIDS Soc. 2019 Jul;22 Suppl 4(Suppl Suppl 4):e25298. doi: 10.1002/jia2.25298. PMID 31328444
- [Background] Celum, C., et al. Risk behavior, perception, and reasons for PrEP among young African women in HPTN 082. in Conference on Retroviruses and Opportunistic Infections.
- [Background] Price JT, Rosenberg NE, Vansia D, Phanga T, Bhushan NL, Maseko B, Brar SK, Hosseinipour MC, Tang JH, Bekker LG, Pettifor A. Predictors of HIV, HIV Risk Perception, and HIV Worry Among Adolescent Girls and Young Women in Lilongwe, Malawi. J Acquir Immune Defic Syndr. 2018 Jan 1;77(1):53-63. doi: 10.1097/QAI.0000000000001567. PMID 28991885
- [Background] Ajayi AI, Mudefi E, Yusuf MS, Adeniyi OV, Rala N, Goon DT. Low awareness and use of pre-exposure prophylaxis among adolescents and young adults in high HIV and sexual violence prevalence settings. Medicine (Baltimore). 2019 Oct;98(43):e17716. doi: 10.1097/MD.0000000000017716. PMID 31651904
- [Background] Muwonge TR, Nsubuga R, Brown C, Nakyanzi A, Bagaya M, Bambia F, Katabira E, Kyambadde P, Baeten JM, Heffron R, Celum C, Mujugira A, Haberer JE. Knowledge and barriers of PrEP delivery among diverse groups of potential PrEP users in Central Uganda. PLoS One. 2020 Oct 28;15(10):e0241399. doi: 10.1371/journal.pone.0241399. eCollection 2020. PMID 33112907
- [Background] Uganda AIDS Commission, The National HIV and AIDS Research Agenda for 2020/21-2024/25. 2021.
- [Background] Albert D, Chein J, Steinberg L. Peer Influences on Adolescent Decision Making. Curr Dir Psychol Sci. 2013 Apr;22(2):114-120. doi: 10.1177/0963721412471347. PMID 25544805
- [Background] Brown, B.B. and J. Larson, Peer relationships in adolescence. 2
- [Background] Ciranka S, van den Bos W. Social Influence in Adolescent Decision-Making: A Formal Framework. Front Psychol. 2019 Aug 29;10:1915. doi: 10.3389/fpsyg.2019.01915. eCollection 2019. PMID 31555164
- [Background] Ndhlovu CE, Kouamou V, Nyamayaro P, Dougherty L, Willis N, Ojikutu BO, Makadzange AT. The transient effect of a peer support intervention to improve adherence among adolescents and young adults failing antiretroviral therapy in Harare, Zimbabwe: a randomized control trial. AIDS Res Ther. 2021 Jun 16;18(1):32. doi: 10.1186/s12981-021-00356-w. PMID 34134738
- [Background] Bakesiima R, Beyeza-Kashesya J, Tumwine JK, Chalo RN, Gemzell-Danielsson K, Cleeve A, Larsson EC. Effect of peer counselling on acceptance of modern contraceptives among female refugee adolescents in northern Uganda: A randomised controlled trial. PLoS One. 2021 Sep 2;16(9):e0256479. doi: 10.1371/journal.pone.0256479. eCollection 2021. PMID 34473750
- [Background] Flanagan S, Gorstein A, Nicholson M, Bradish S, Amanyire D, Gidudu A, Aucur F, Twesigye J, Kyateka F, Balamaga S, Buttenheim A, Zimmerman E. Behavioural intervention for adolescent uptake of family planning: a randomized controlled trial, Uganda. Bull World Health Organ. 2021 Nov 1;99(11):795-804. doi: 10.2471/BLT.20.285339. Epub 2021 Sep 29. PMID 34737472
- [Background] Tapera T, Willis N, Madzeke K, Napei T, Mawodzeke M, Chamoko S, Mutsinze A, Zvirawa T, Dupwa B, Mangombe A, Chimwaza A, Makoni TM, Mandewo W, Senkoro M, Owiti P, Tripathy JP, Kumar AMV. Effects of a Peer-Led Intervention on HIV Care Continuum Outcomes Among Contacts of Children, Adolescents, and Young Adults Living With HIV in Zimbabwe. Glob Health Sci Pract. 2019 Dec 23;7(4):575-584. doi: 10.9745/GHSP-D-19-00210. Print 2019 Dec 23. PMID 31852741
- [Background] International HIV/AIDS Alliance, Supporting children, adolescents and young people living with HIV to start and stay on HIV treatment.